CLINICAL TRIAL: NCT02532933
Title: Influence of Patellar Geometry on Kinematics, Quadriceps Function, and Patient Outcome in Subjects With the Attune PS RP
Brief Title: Stereo Radiography of TKA Patella Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: DePuy Synthes (Industry); Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Kevin Shelburne, Senior Research Engineer, University of Denver
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 779383 2015 Attune Patella
Record Dates: First submitted 2015-08-18; First posted 2015-08-26 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Total Knee Arthroplasty
Keywords: Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medialized Dome Patella (Active Comparator): Subjects with total knee arthroplasty using the DePuy Synthes Attune Posterior Stabilized Rotating Platform including patella resurfacing with a medialized dome component geometry
  Interventions: Device: DePuy Synthes Attune PS RP
- Anatomic Patella (Active Comparator): Subjects with total knee arthroplasty using the DePuy Synthes Attune Posterior Stabilized Rotating Platform including patella resurfacing with an anatomic component geometry
  Interventions: Device: DePuy Synthes Attune PS RP

INTERVENTIONS:
Device: DePuy Synthes Attune PS RP

SUMMARY:
The overall purpose is to compare the kinematics and mechanics of medialized dome and anatomic resurfacing through measurement and simulation, and to correlate these findings with patient satisfaction and performance.

Aim 1: Comparison of patellofemoral kinematics between dome and anatomic implant designs using stereo radiography and correlation with patient function as measured by Knee injury and Osteoarthritis Outcome score, Knee Society score, and strength.

Hypothesis: the anatomic patellar implant will have significantly greater sagittal flexion than the dome implant.

Aim 2: Comparison of dome and anatomic moment arm, quadriceps efficiency, patellar contact mechanics and loading through the use of subject-specific simulation.

Hypothesis: quadriceps efficiency and moment arm will be greater for the anatomic patellar implant, while loading between the patellar and femoral components will be reduced.

DETAILED DESCRIPTION:
Successful function and outcome following total knee arthroplasty (TKA) is partly determined by the restoration of patellofemoral (PF) function and recovery of the quadriceps mechanism of the knee. Patients with TKA often exhibit adaptations in their movement patterns during functional activity that have been attributed to quadriceps strength reduction and activation deficits that may be linked to the mechanics of the reconstructed knee. Changes in the articular geometry with patella resurfacing also affect patellofemoral kinematics, contact mechanics and loading on the patellar bone. While movement adaptations persist in patients with TKA long after knee repair, measurement of the 6 degree-of-freedom (DOF) kinematics of the patellofemoral joint are difficult with traditional motion capture methods. High-speed stereo radiography (HSSR), an advancement of biplane fluoroscopy, enables measurement of bone and implant motion during activity with sub-mm accuracy. The ability to measure and model the kinematics of the knee with this precision can improve understanding of implanted knee mechanics. What's more, acquiring HSSR in synchrony with whole-body measurements (body segment video motion capture, muscle electromyography (EMG), and ground forces) establishes connections between joint-level and whole-body function, and enables creation of subject-specific models of the knee and lower extremity. Integration with modeling is important because it reveals the biomechanical consequences of differences in patellofemoral kinematics.

Previous measurement and modeling comparisons of PF kinematics between dome and anatomic resurfacing designs have revealed differences in patellar sagittal plane flexion that have implications for quadriceps efficiency and patient satisfaction. Quadriceps efficiency is a measure of the effective moment arm of the quadriceps muscles; greater efficiency allows the quadriceps to produce knee extensor torque with less force. Patellar flexion can alter quadriceps efficiency by changing the moment arm of the patellar tendon and the way the patella transmits quadriceps force due to changes in patellofemoral contact. Patient satisfaction may be affected by changes in quadriceps efficiency through increased extensor mechanism strain and changes in load transfer that may be linked to anterior knee pain. While HSSR measurements can elucidate differences in dome and anatomic kinematics, computational modeling is required to determine how kinematic differences affect joint and muscle forces and overall limb functionality.

Aim 1: Comparison of patellofemoral kinematics between dome and anatomic implant designs using stereo radiography and correlation with patient function as measured by Knee injury and Osteoarthritis Outcome score, Knee Society score, and strength. Laboratory measurements will be collected from 22 TKA patients with medialized dome and 22 TKA patients with medialized anatomic patellae. Equal numbers of men and women will be recruited for the study. The angle of the patellar component relative to the femoral component will be measured and compared to reported values in healthy subjects. Correlations will be made with patient outcome scores.

Aim 2: Comparison of dome and anatomic moment arm, quadriceps efficiency, patellar contact mechanics and loading through the use of subject-specific simulation. Moment arm will be measured in millimeters as the distance from the patellar tendon to the knee joint center of rotation, and compared to values reported for the healthy knee. Quadriceps efficiency will be calculated as the ratio of quadriceps force to patellar tendon force. Patellar contact mechanics are defined as the force and location of force between the patellar and femoral components.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Age: 18-80 years
* Unilateral or bilateral total knee replacement with an Attune posterior-stabilized rotating-platform implant including either medialized dome or medialized anatomic patellae
* Minimum 9 months post TKA procedure

Exclusion Criteria:

* Concomitant lower extremity injury that continues to cause pain or loss of normal function (70 or greater Knee Society score)
* Inactive or unable to participate for health reasons (40 or greater on the physical component scale and and the mental component scale composite scores of the SF-12 Health Survey)
* Neurologic deficit that affects function or understanding of testing protocol
* Pregnant
* Other participation in a research study involving exposure to x-ray radiation
* body mass index greater than 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shelburne, PhD, Principal Investigator — University of Denver

REFERENCES:
- See also: Website of the Center for Orthopaedic Biomechanics — http://www.du.edu/biomechanics

RESULTS

PARTICIPANT FLOW:
Groups:
- Medialized Dome Patella: Subjects with total knee arthroplasty using the DePuy Synthes Attune Posterior Stabilized Rotating Platform including patella resurfacing with a medialized dome component geometry
  DePuy Synthes Attune PS RP
- Anatomic Patella: Subjects with total knee arthroplasty using the DePuy Synthes Attune Posterior Stabilized Rotating Platform including patella resurfacing with an anatomic component geometry
  DePuy Synthes Attune PS RP
Period: Overall Study
Arm/Group | Medialized Dome Patella | Anatomic Patella
Started | 22 | 22
Completed | 16 | 16
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medialized Dome Patella | Anatomic Patella | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (5.3) | 65.2 (6.8) | 63.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Patellar Flexion Measured as the Relative Angle Between the Femoral and Patellar Components of the Implant.
Description: Difference between dome and anatomic patellofemoral flexion, which is measured as the relative angle between the femoral and patellar components of the implant.
Time Frame: One day
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Medialized Dome Patella | Anatomic Patella
Number analyzed (Participants) | 16 | 16
degrees | 29.6 (8.1) | 21.0 (6.7)

ADVERSE EVENTS:
Time Frame: 2 to 3 hours
Description: Data was collected in a human motion laboratory on one day for each participant. An adverse event was defined as any adverse occurrence during the 2 to 3 hour data collection
Arm/Group | Medialized Dome Patella | Anatomic Patella
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT02532933/Prot_SAP_000.pdf